CLINICAL TRIAL: NCT07138404
Title: Assessment of Psychological Stress Among Dental Students During Clinical Training at Cairo University: A Cross-Sectional Study
Brief Title: STRESS AMONG DENTAL STUDENT DURING DENTAL TRAINING
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, MOUAWIA AHMAD ABLA, RESEAECH CANDIDTE, Cairo University
Other Study IDs: 3111998
Record Dates: First submitted 2025-07-01; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Stress Among Dental Students

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dental student: dental student in year 4 and year 5 practicing dental procedure in conservative and endodontics department
  Interventions: Other: self administration questioner

INTERVENTIONS:
Other: self administration questioner — A self questionnaire will be distributed to evaluate the levels of stress experienced by dental students currently undertaking clinical training in 4th and 5th academic years at Cairo University during the performance of specific clinical procedures in conservative and endodontics treatment.The data obtained from the questionnaire will be statistically analyzed to identify and interpret the variations in the results.

SUMMARY:
A self questionnaire will be distributed to evaluate the levels of stress experienced by dental students currently undertaking clinical training in 4th and 5th academic years at Cairo University during the performance of specific clinical procedures in conservative and endodontics treatment.The data obtained from the questionnaire will be statistically analyzed to identify and interpret the variations in the results.

ELIGIBILITY:
Inclusion Criteria:

- 1)Undergraduate dental students officially enrolled at Cairo University. 2)Students currently undertaking clinical training, (e.g., 4th and 5th academic years) 3)Students who have participated in clinical procedures such as restorative treatments and root canal therapy.

4)Students aged between 20 and 25 years Willingness to participate and provide informed consent electronically.

Exclusion Criteria:

* 1)Pre-clinical dental students (1st to 3rd academic years) who have not yet begun clinical exposure.

  2)Students who are not actively enrolled during the study period or are on academic leave.

  3)Responses that are incomplete or missing key sections of the questionnaire. Recent graduates or individuals are no longer engaged in the undergraduate academic program.

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: dental in year4 and year 5 in Cairo university practicing dental procedure in conservative and endodontics departments.
Sampling Method: Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of stress among dental students | up to 24 week
  Prevalence of stress among dental students in year 4 and year 5 practicing dental procedure in conservative and endodontics department

IPD SHARING:
Plan to Share IPD: Undecided